CLINICAL TRIAL: NCT00470392
Title: Mechanistically-based Optimization of UV Radiation Therapy in Psoriasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting complete and administrative termination
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single
Other Study IDs: IMMB-004-06S
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis
Keywords: Erythema; optimization; Papule; Plaque; pretreatment; T cells; UVB laser light; psoriasis; topical administration
MeSH Terms: conditions — Psoriasis; Erythema; Plaque, Amyloid | interventions — Imiquimod; Clobetasol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imiquimod (Other): Each study subject served as his/her own control. For this arm of the study, topical vehicle was applied to one plaque for 5 days. Imiquimod (5% topical cream) was applied to two psoriasis plaques for 5 days. Skin biopsies were taken from half of each of the 3 plaques at specific time points after completion of topical pre-treatment. The other half of the plaques were exposed to UVB light (via Excimer laser). Biopsies were subsequently taken at a specified time point.
  Interventions: Drug: Imiquimod
- Clobetasol (Other): Each study subject served as his/her own control. For this arm of the study, topical vehicle was applied to one plaque for 5 days. Clobetasol propionate 0.05% was applied to two psoriasis plaques for 5 days. Skin biopsies were taken from half of each of the 3 plaques at specific time points after completion of topical pre-treatment. The other half of the plaques were exposed to UVB light (via Excimer laser). Biopsies were subsequently taken at a specified time point.
  Interventions: Drug: Clobetasol

INTERVENTIONS:
Drug: Imiquimod — Each study subject served as his/her own control. For this arm of the study, topical vehicle was applied to one plaque for 5 days. Imiquimod (5% topical cream) was applied to two psoriasis plaques for 5 days. Skin biopsies were taken from half of each of the 3 plaques at specific time points after completion of topical pre-treatment. The other half of the plaques were exposed to UVB light (via Excimer laser). Biopsies were subsequently taken at a specified time point.
  Other Names: Aldara
  Arms: Imiquimod
Drug: Clobetasol — Each study subject served as his/her own control. For this arm of the study, topical vehicle was applied to one plaque for 5 days. Clobetasol propionate 0.05% was applied to two psoriasis plaques for 5 days. Skin biopsies were taken from half of each of the 3 plaques at specific time points after completion of topical pre-treatment. The other half of the plaques were exposed to UVB light (via Excimer laser). Biopsies were subsequently taken at a specified time point.
  Other Names: Temovate
  Arms: Clobetasol

SUMMARY:
The purpose of this study is 1) to determine whether Imiquimod or Steroid pretreatment modifies UVB laser light response resulting in increased cell death compared to UVB laser light alone; 2) to determine if pretreatment of psoriatic lesions with Imiquimod or Steroid prior to UVB laser light exposure selectively effects various T cell functions; 3) to determine clinical results from the Imiquimod/Steroid/UVB laser light and correlate those changes with immuno-histochemical changes in the skin; and 4) to determine if single high dose lesion limited UVB laser light intervention combined with Imiquimod or Steroid influences T cell changes

DETAILED DESCRIPTION:
The characteristic lesion of psoriasis is a sharply demarcated erythematous papule or plaque with excessive scaling due to hyperproliferating keratinocytes, infiltrating granulocytes, and a dense mononuclear infiltrate with activated T cells. To date, no one mechanism has been explanatory for the panoply of changes that occur in both the dermis and epidermis of psoriasis patients. Several key findings have shown that cutaneous T cells play a key role in the propagation of the disease; memory-type T cells home to the skin, specifically due to expression of cutaneous lymphocyte antigen (CLA), and are the main effector cells in psoriatic tissue responsible for the production of cytokines that result in exacerbated cutaneous inflammation. T cell recruitment is thought to occur in psoriasis, in part, as a result of cytokine and chemokine release from keratinocytes, macrophages, and endothelial cells. CLA-positive T cells migrate into the tissues where memory-effector T cells are activated and expand. This migration is critical to maintenance of the psoriasis lesions, because anti-LFA-1 antibodies (efalizumab) are effective in treating psoriasis, resulting in blood lymphocytosis and tissue depletion of T cells. Despite many years of using UVB phototherapy in the treatment of psoriasis, its mechanism of action is based mainly on in vitro exposures of isolated cells and on extrapolations from UV effects on normal skin, with little direct data from lesional skin.

Previously, our studies determined optimal single efficacious dose using the Excimer laser, refined the mechanism of UVB action in psoriasis, developed key cytokine quantitative meth -ods to assess targeted mRNA levels in psoriatic tissue after treatment, demonstrated that regulatory T cells from psoriasis tissue and blood appear to have a functional defect, and demonstrated that UVA component of solar radiation is a critical and significant contributor to UV-induced in vivo immuno-suppression. All of these previous findings lead us to our current hypothesis that direct selective apoptotic effects on the T mem/Teff cells may result in decreased APC activation and IL-12 over-riding of Treg suppression and a re-balanced Tre:Tmem/eff cell ratio which in turn may have a sustained remittive effect (high duration multi-month clearing of a psoriasis lesion after a single UVB laser light treatment.)

ELIGIBILITY:
Inclusion Criteria:

* The presence of plaque-type psoriasis in areas of the trunk, buttocks, or extremities that are amenable to biopsy and evaluable disease in at least 2 cm target treatment sites separated by 1 cm
* Age 18-80, both genders, all ethnicities
* No contraindications to phototherapy or biopsy procedures
* No topical steroid, tar, phototherapy, Vitamin D, or retinoid therapy to target lesions for at least 1 week prior to the study
* No systemic psoriasis therapy for at least four weeks prior to the study
* Able to give informed consent under IRB approval procedures

Exclusion Criteria:

* Photosensitivity disorders
* Active untreated diseases or medication usage which may interfere with UVB, wound healing, or immune function
* Hypersensitivity to local anesthetic
* Inability to provide informed consent
* Pregnancy and /or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cooper, MD, Principal Investigator — VA Medical Center-Cleveland
Locations (2):
- United States (2):
  - University Hospital Case Medical Center, Cleveland, Ohio
  - VA Medical Center, Cleveland, Cleveland, Ohio

REFERENCES:
- See also: The National Institute of Arthritis, Musculoskeletal, and Skin Diseases website providing fast facts on health topics, including psoriasis — http://www.niams.nih.gov/Health_Info/psoriasis/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Dermatology clinics at University Hospitals Case Medical Center and the Louis Stokes Cleveland VAMC.
Pre-assignment Details: Subjects with moderate to severe psoriasis were recruited from May 2007 to July 2012. 23 subjects were screened but only 9 were assigned to a study arm and received treatment. Per protocol, subjects underwent a washout period of 1 week for topical treatments and 1 month for systemic treatments prior to pre-treatment with Imiquimod or Clobetasol.
Period: Overall Study
Arm/Group | Imiquimod | Clobetasol
Started | 7 (Number of subjects enrolled, passed screening and assigned to this arm.) | 2 (Number of subjects enrolled, passed screening and assigned to this arm.)
Completed | 7 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imiquimod | Clobetasol | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 80 years | 7 | 2 | 9
  >=80 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Elevated MyxA
Description: Lesions were treated with either Imiquimod or Clobetasol cream. Lesions were subsequently treated with UVB and biopsied. From the biopsy samples obtained from the Imiquimod arm, quantitative PCR was performed to measure levels of Myx A, an imiquimod response gene.
Time Frame: Biopsy samples for analysis were taken 1 hour post UVB treatment
Population: Per protocol.
Measure: Number; unit: participants
Groups:
- Clobetasol: Each study subject served as his/her own control. For this arm of the study, topical vehicle was applied to one plaque for 5 days. Clobetasol propionate 0.05% was applied to two psoriasis plaques for 5 days. Skin biopsies were taken from half of each of the 3 plaques at specific time points after completion of topical pre-treatment. The other half of the plaques were exposed to UVB light (via Excimer laser). Biopsies were subsequently taken at a specified time point. No synchronized T cell reactivation was observed upon immunohistochemical analysis, nor upon analysis of T cell death associated gene (TDAG) mRNA by PCR, with Clobetasol treatment, so this arm was terminated.
Arm/Group | Imiquimod | Clobetasol
Number analyzed (Participants) | 7 | 0
participants | 1 |

2. Secondary Outcome: Number of Subjects With Improvement in Lesional Psoriasis Area and Assessment (PASI) Score After Imiquimod and UVB Treatment
Description: The PASI is a disease burden measure that integrates area, erythema, thickness and scale of each target lesion. The severity score for each region is calculated by adding the scores for redness, thickness and scale (each of which are graded from 0 to 4). The maximum severity score is 12. The higher the PASI, the worse the disease. Thus, an improvement in PASI score is a lower score than the pre-treatment PASI.
Time Frame: 2 weeks after Imiquimod and UVB
Population: Per protocol.
Measure: Number; unit: participants
Arm/Group | Imiquimod | Clobetasol
Number analyzed (Participants) | 7 | 0
participants | 4 |

3. Secondary Outcome: Number of Subjects With a 1.5 Fold Increase in mRNA Expression of GRAMD1A and DMXL2
Description: Based upon upregulated mRNA expression of MyxA in 1 out of 7 patients treated with Imiquimod, a list of alternative target genes responsive to Imiquimod was generated. The target mRNAs examined included GRAMD1A, IL2RA, TGHD1, DMXL2. The target gene was consider upregulated if there was a 1.5 fold increase in the mRNA expression of the target gene.
Time Frame: Biopsy samples for analysis were taken 1 hour post UVB treatment
Measure: Number; unit: participants
Arm/Group | Imiquimod | Clobetasol
Number analyzed (Participants) | 7 | 0
participants | 1 |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 30 days. The investigators assessed for adverse events at each study visit.
Arm/Group | Imiquimod | Clobetasol
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 4/7 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod (N=7) | Clobetasol (N=2)
Exacerbation of non-target psoriasis plaques during washout of topical medications (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Grade 4 target site reaction - blistering post UVB (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Common cold (Infections and infestations) | 0 (0) | 1 (1)
Contact vs irritant dermatitis surrounding target sites secondary to bandages (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Grade 3 target site reaction - erythema with mild discomfort post UVB (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Exacerbation of psoriasis surrounding target sites secondary to bandages (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (General disorders) | 0 (0) | 1 (1) — evaluated and treated by the staff of the LSCVAMC Emergency Department
Burning sensation with use of study product (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Right knee trauma and pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No synchronized T cell reactivation was observed upon immunohistochemical analysis, nor upon analysis of T cell death associated gene (TDAG) mRNA by PCR, with Clobetasol treatment, so this arm was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No